CLINICAL TRIAL: NCT00864318
Title: Dose Intensification Phase II Study in Refractory Germ Cell Tumors With Relapse and Bad Prognosis. TICE Protocol : Paclitaxel and Ifosfamide Followed by Carboplatine and Etoposide Intensification With Individual Carboplatine Dose Adjustment.
Brief Title: Dose Intensification Study in Refractory Germ Cell Tumors With Relapse and Bad Prognosis
Acronym: TICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08 GENH 06
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Germ Cell Tumors
Keywords: refractory; germ cell tumors; relapse; bad prognosis; Refractory germ cell tumors with relapse and bad prognosis
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Recurrence | interventions — Paclitaxel; Ifosfamide; Carboplatin; Etoposide; Cytapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paclitaxel — 200mg/m2 for 3 hours at Cycle 1 day 1 and Cycle 2 day 1 with 14 days between cycles
  Other Names: Taxol
Drug: Ifosfamide — 2g/m²/day in 1 liter of G5 for 3 hours at Cycle 1 and Cycle 2 from day 2 to day 4 with 14 days between cycles
  Other Names: Holoxan
Drug: Carboplatine — From cycle 3 to cycle 5 :
  Carboplatine is administered with AUC = 24 mg/mL x min from Day 1 to Day 3. Day 3 Carboplatine dose is calculated taking into account real creatinine clearance defined at day 1 for each patient
Drug: Etoposide — From Cycle 3 to cycle 5, 400mg/m2/day from day 1 to day 3
  Other Names: VP16
Procedure: cytapheresis + transfusion of autologous peripheral blood stem cells — Cytapheresis occured between day 11 and day 13 of the 2 first cycle (Taxol® +Holoxan®). Cytapheresis total objective is 9X106 CD34+/kg of patient weight.
  At cycle 3, 4 and 5 at day 5 : Re-injection of stem cells (1/3 with minimum 2.106 CD34/kg) 48 hours after chemotherapy end

SUMMARY:
Not randomized, multicentric, national phase II trial estimating the efficacy of an intensification protocol in patients with refractory germ cell tumors with relapse and bad prognosis.

Treatment consists in two Paclitaxel and Ifosfamide intensification cycles followed by three Carboplatine and Etoposide high dose cycles. The point is the individual Carboplatine adjustment to take into account inter-individual patients variability.

This adaptation allow to control each patient plasmatic exposition to avoid both inacceptable toxicities (such as ear toxicity) and a low exposition losing then the benefit of this high dose protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Germ cell tumors whatever histology (TGNS or séminoma : TGS ) whose origin is gonadic, extra-gonadic, retro-peritoneal or primitive mediastinal
2. Age >= 18 years old
3. Histologically confirmed germ cell tumor (TGS) or biomarkers rate allowing to diagnose germ cell tumor without histology (TGNS)
4. Relapse or progression with bad prognosis in 1st treatment line : One of these criteria valid point 4 :

   progression after incomplete clinical response (Stable disease) to a Cisplatin basis chemotherapy; biomarker progression 4 weeks following the last chemotherapy cycle administration; progression during the first treatment line without obtention of at least stable disease; primitive mediastinal origin in first relapse.
5. TGNS or TGS in relapse after 2 treatment lines
6. Disease progression ( previous points 4 or 5) documented by :

   tumors biomarkers increase (AFP and/or HCG) if no, a biopsy is needed to confirm presence of tumors active cells
7. ECOG Performance status 0-2
8. Biological Function :

   Neutrophils >= 1500/mm3, Platelets >= 150.000/mm3 ; normal creatinine (or clearance >= 50 ml/mn) ; SGOT, SGPT <= 2,5N (or 5N if hepatic metastases), Bilirubin < 1,5N
9. Cardiac Functions (FEV >= 50%), Respiratory Functions , neurological Functions compatibles with high dose chemotherapy administration
10. Absence of previous intensification
11. Patient Information and Informed consent signature
12. HIV and B and C hepatitis negative serologies
13. Negative pregnancy test for women with reproductive potential and adequate contraception before study entry
14. Patient affiliated to social security system

Exclusion Criteria:

1. Patients whose diagnosis of relapse was not confirmed by an anatomopathological examination or by an increase of tumors markers
2. Primitive encephalic germ cell tumors
3. Germ cell tumors in relapse with favorable factors of treatment response to conventional chemotherapy (RC sustainable after Cisplatin): prior cRC or incomplete clinical response but with normalization of markers and testicular origin
4. Growing Teratoma lesions
5. Patients with HIV infection, hepatitis B and C
6. Patients with symptomatic brain metastases despite appropriate corticosteroid treatment
7. Associated pathology may prevent the patient to receive treatment, creatinine clearance ≤ 50 mL / min (calculated by Cockcroft-Gault)
8. FEV <50%
9. History of cancer (except basal cell epithelioma skin cancer) in the 3 years preceding the entry into the trial
10. Patient already included in another clinical trial involving an experimental molecule
11. Pregnant or breast feeding women
12. Persons without liberty or under guardianship,
13. Geographical, social or psychological conditions that do not permit compliance with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-03-13 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Complete response rate(by chemotherapy or chemotherapy + surgery), pathological complete response rate. | 6 months

SECONDARY OUTCOMES:
Progression free survival | 8 years
Time to progression | 8 years
Toxicity | 6 months
To find a predictive value for Cystatin C as a biomarker of renal function to avoid next to follow plasmatic concentrations to adapt Carboplatine dose in TICE protocol. | 4 years
Etoposide pharmacokinetics (in particular inter-individual variability of Etoposide plasmatic concentrations AUC in such patients | 4 years
Genetic polymorphisms involved in response and safety treatments | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHEVREAU, MD, Principal Investigator — Institut Claudius Regaud
Locations (12):
- France (12):
  - Centre Paul Papin, Angers
  - Hopital St André, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHU, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut Val d'aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital TENON, Paris
  - CHU, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Chevreau C, Massard C, Flechon A, Delva R, Gravis G, Lotz JP, Bay JO, Gross-Goupil M, Fizazi K, Mourey L, Paci A, Guitton J, Thomas F, Lelievre B, Ciccolini J, Moeung S, Gallois Y, Olivier P, Culine S, Filleron T, Chatelut E. Multicentric phase II trial of TI-CE high-dose chemotherapy with therapeutic drug monitoring of carboplatin in patients with relapsed advanced germ cell tumors. Cancer Med. 2021 Apr;10(7):2250-2258. doi: 10.1002/cam4.3687. Epub 2021 Mar 5. PMID 33675184